CLINICAL TRIAL: NCT03556033
Title: Effect of the SGLT-2 Inhibitor Dapagliflozin on Impaired Awareness of Hypoglycemia in Type 1 Diabetes
Brief Title: Effect of Dapagliflozin on IAH in T1DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T1DM_IAH_dapa
Record Dates: First submitted 2018-05-17; First posted 2018-06-14 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia; Hypoglycemia Unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin 10 mg capsule once daily for 8 weeks
  Interventions: Drug: Dapagliflozin
- Placebo oral capsule (Placebo Comparator): Placebo matched to dapagliflozin 10 mg capsule once daily for 8 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Dapagliflozin — 8 weeks treatment with dapagliflozin on top of insulin treatment
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo oral capsule — 8 weeks treatment with placebo capsules on top of insulin treatment
  Arms: Placebo oral capsule

SUMMARY:
Approximately 25% of patients with type 1 diabetes have lost the capacity to timely detect hypoglycaemia, a condition referred to as impaired awareness of hypoglycaemia (IAH) that causes a six-fold higher risk of severe, potentially hazardous, hypoglycaemia. IAH is usually the end-result of a process of habituation to recurrent hypoglycaemia that is potentially reversible. Treatment with sodium glucose cotransporter (SGLT)-2 inhibitors (SGLT-2i) in addition to insulin therapy may decrease the incidence of hypoglycaemia in patients with type 1 diabetes. This study will test the hypothesis that treatment with the SGLT-2 inhibitor, dapagliflozin, added to basal-bolus insulin therapy will improve awareness of hypoglycaemia in patients with type 1 diabetes and IAH. In a randomized doubleblind placebo-controlled cross-over trial, patients will be treated for 8 weeks with dapagliflozin (or placebo), after which hypoglycemic symptoms and counterregulatory hormone responses will be examined during a hyperinsulinemic hypoglycemic glucose clamp study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, disease duration >1 year
* Age >18 years, <75 years
* BMI 19-40 kg/m^2
* Insulin treatment according to basal-bolus insulin regimen (injections or insulin pump)
* Impaired awareness of hypoglycemia as assessed by a score of 3 or more on the modified Dutch translation of the Clarke questionnaire
* Glycated haemoglobin (HbA1c) ≥42 mmol/mol (6%) and ≤75 mmol/mol (9.0%)
* Ability to provide informed consent

Exclusion Criteria:

* Treatment with SGLT-2 inhibitors
* Known intolerance to SGLT-2 inhibitors
* Treatment with loop diuretics or other anti-hypertensive agents
* Treatment with glucose-modifying (other than insulin) or immune-modifying agents (e.g. prednisolon)
* Treatment with pioglitazone
* Use of statins
* A history of cardiovascular disease (e.g. myocardial infarction, stroke, heart failure) or hypotension
* A history of galactose-intolerance, lactase deficiency, glucose-galactose malabsorption
* History of diabetic ketoacidosis requiring medical intervention within 1 month before screening
* Admission to the hospital for hyperglycemia or hypoglycemia within 1 month before screening
* Frequent episodes of severe hypoglycemia within 1 month before screening
* Laser coagulation for proliferative retinopathy (past 6 months)
* Proliferative retinopathy
* Diabetic nephropathy as reflected by an albumin-creatinin ratio ˃ 30 mmol/mg or an estimated glomerular filtration rate (by MDRD) ˂60ml/min/1.73m2
* History of pancreatitis (acute or chronic) or pancreatic cancer
* Use of premixed insulin or of long-acting insulin alone
* Total daily insulin dose requirements <20 units unless on pump treatment
* Pregnancy or unwillingness to undertake measures for birth control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Symptom score in response to insulin-induced hypoglycaemia | 45 minutes
  Symptom scores (autonomic, neuroglycopenic and general) measured during hyperinsulinemic hypoglycaemic glucose clamps. This questionnaire consists of 18 symptoms, which can be scored between 0 (none) to 6 (severe). Total scores range between 0 and 108, the higher the score, the more symptoms patients have during and after hypoglycemia.

SECONDARY OUTCOMES:
Counterregulatory hormone responses to insulin-induced hypoglycaemia | 45 minutes
  (nor)adrenaline, glucagon, insulin, growth hormone and cortisol responses to hypoglycaemia measured during hyperinsulinemic hypoglycaemic glucose clamps
Time until glycaemic recovery from hypoglycaemia | 45 minutes
  measured during hyperinsulinemic hypoglycaemic glucose clamps
Maximal glucose excursion post-hypoglycaemia | 45 minutes
  Maximal glucose level (mmol/l) measured during the 90 minutes after ending the hypoglycaemic phase of the clamp (during restoration of euglycaemia)
Time until glucose peak post-hypoglycaemia | 45 minutes
  measured during hyperinsulinemic hypoglycaemic glucose clamps
Area under the glucose concentration curve post-hypoglycaemia | 45 minutes
  measured during hyperinsulinemic hypoglycaemic glucose clamps
Number of severe hypoglycaemic events during follow-up | 16 weeks
  measured during follow-up
Number of nocturnal hypoglycaemic events during follow-up | 16 weeks
  measured during follow-up
Number of any hypoglycaemic events during follow-up | 16 weeks
  measured during follow-up
Time spent under hypoglycaemic conditions measured by glucose sensor monitoring | 2 weeks
  measured during follow-up
Glucose variability as measured by glucose sensor monitoring | 2 weeks
  measured during follow-up

OTHER OUTCOMES:
Inflammatory/atherogenic phenotype of circulating monocytes from the participating patients | 45 minutes
  measured during hyperinsulinemic hypoglycaemic glucose clamps

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No